CLINICAL TRIAL: NCT02074982
Title: A 52-week, Multicenter, Randomized, Double-blind Study of Subcutaneous Secukinumab to Demonstrate Efficacy as Assessed by Psoriasis Area and Severity Index at 16 Weeks of Treatment Compared to Ustekinumab and to Assess Long-term Safety, Tolerability and Efficacy in Subjects With Moderate to Severe Plaque Psoriasis (CLEAR)
Brief Title: Efficacy of Secukinumab Compared to Ustekinumab in Patients With Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2317; 2013-003434-32 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Chronic Plaque Type Psoriasis
Keywords: chronic plaque type psoriasis, secukinumab, ustekinumab, inflammatory skin disease, scaling
MeSH Terms: conditions — Dermatitis | interventions — secukinumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AIN457 300 mg (Experimental): patients received AIN457 (secukinumab) 300 mg (two secukinumab 150 mg injections) s.c. (subcutaneously) once every week at weeks 0, 1,2,3, followed by monthly dosing starting at week 4 to week 48 inclusive
  Interventions: Drug: AIN457 300 mg
- Ustekinumab (Active Comparator): patients received ustekinumab 45/90 mg (weight depended, according to label) s.c. (subcutaneously) and/or placebo secukinumab injections once every week at weeks 0,1,2, and 3 followed by monthly dosing starting at week 4 to week 48 inclusive
  Interventions: Drug: ustekinumab 45/90 mg; Drug: placebo secukinumab

INTERVENTIONS:
Drug: AIN457 300 mg
  Other Names: secukinumab
  Arms: AIN457 300 mg
Drug: ustekinumab 45/90 mg
  Arms: Ustekinumab
Drug: placebo secukinumab — Placebo
  Arms: Ustekinumab

SUMMARY:
This study assessed efficacy of secukinumab, compared to ustekinumab, in patients that have plaque-type psoriasis

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe plaque type psoriasis for at least 6 months before randomization
* patients eligible for systemic therapy with inadequately controlled psoriasis

Exclusion Criteria:

* forms of sporiasis other than plaque type psoriasis
* previous exposure to secukinumab, ustekinumab, or other biologic drugs targeting (IL)-17A or IL-17RA

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (119):
- United States (25):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Arlington Heights, Illinois
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Forest Hills, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Australia (4):
  - Novartis Investigative Site, Phillip, Australian Capital Territory
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
- Austria (3):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (4):
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Novartis Investigative Site, Arhus C, Denmark
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
- Germany (17):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Pommelsbrunn
- Novartis Investigative Site, Heraklion, Crete, GR, Greece
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Verona, VR
- Netherlands (5):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, Zwijndrecht
- Novartis Investigative Site, Bergen, Norway
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Slovakia (4):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Kosice-Saca, Slovak Republic
  - Novartis Investigative Site, Bojnice
  - Novartis Investigative Site, Košice
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Gwangju
- Spain (15):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lausanne, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Bursa
- United Kingdom (8):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Redhill, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Alpalhao M, Duarte J, Diogo R, Vandemeulebroecke M, Ortmann CE, Kasparek T, Filipe P. Lower Limbs are the Most Difficult-to-Treat Body Region of Patients with Psoriasis: Pooled Analysis of CLEAR and CLARITY Studies of Secukinumab Versus Ustekinumab by Body Region. BioDrugs. 2022 Nov;36(6):781-789. doi: 10.1007/s40259-022-00558-2. Epub 2022 Nov 5. PMID 36334236
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Conrad C, Ortmann CE, Vandemeulebroecke M, Kasparek T, Reich K. Nail Involvement as a Predictor of Differential Treatment Effects of Secukinumab Versus Ustekinumab in Patients with Moderate to Severe Psoriasis. Dermatol Ther (Heidelb). 2022 Jan;12(1):233-241. doi: 10.1007/s13555-021-00654-1. Epub 2021 Dec 6. PMID 34870789
- [Derived] Augustin M, Thaci D, Eyerich K, Pinter A, Radtke M, Lauffer F, Mrowietz U, Gerdes S, Pariser D, Lebwohl M, Sieder C, Melzer N, Reich K. Continued treatment with secukinumab is associated with high retention or regain of response. Br J Dermatol. 2020 Jan;182(1):67-75. doi: 10.1111/bjd.17991. Epub 2019 Jul 17. PMID 30972746
- [Derived] Thaci D, Blauvelt A, Reich K, Tsai TF, Vanaclocha F, Kingo K, Ziv M, Pinter A, Hugot S, You R, Milutinovic M. Secukinumab is superior to ustekinumab in clearing skin of subjects with moderate to severe plaque psoriasis: CLEAR, a randomized controlled trial. J Am Acad Dermatol. 2015 Sep;73(3):400-9. doi: 10.1016/j.jaad.2015.05.013. Epub 2015 Jun 17. PMID 26092291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 676 patients who were randomized to the study, 571 patients completed the study (286 patients (84.9%) in the secukinumab group and 285 patients (84.1%) in the ustekinumab group. Efficacy Data up to 52 weeks and Safety Data included up to 104 weeks
Period: Overall Study
Arm/Group | AIN457 300 mg | Ustekinumab
Started | 337 | 339
Full Analysis Set (FAS) | 336 | 339
Safety Set (SF) | 335 | 336
Completed | 286 | 285
Not Completed | 51 | 54
Not completed — Adverse Event | 15 | 7
Not completed — Lack of Efficacy | 6 | 1
Not completed — Lost to Follow-up | 9 | 10
Not completed — Non-compliance with study treatment | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 1 | 2
Not completed — Protocol deviation | 4 | 3
Not completed — Technical problems | 0 | 2
Not completed — Subject/guardian decision | 15 | 24
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 300 mg | Ustekinumab | Total
Number analyzed (Participants) | 337 | 339 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.95) | 44.6 (13.67) | 44.9 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 87 | 195
  Male | 229 | 252 | 481

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Moderate to Severe Plaque Psoriasis Who Achieved Psoriasis Area and Severity Index (PASI) 90 at Week 16
Description: Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 90 responders were defined as participants achieving ≥ 90% improvement at Week 16
Time Frame: Week 16
Population: Full Analysis Set (FAS) included all randomized patient minus 1 patient that was excluded due to missing informed consent prior to initiating study procedures.
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 300 mg | Ustekinumab
Number analyzed (Participants) | 334 | 335
Percentage of Participants | 79.0 | 57.3
Statistical Analysis 1: Comparison: AIN457 300 mg vs Ustekinumab; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.85, 95% CI 2-sided [2.01 to 4.02]

2. Secondary Outcome: Speed of Onset Based on the Percentage of Participents Achieving PASI 75 at Week 4
Description: Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  Speed of Onset was based on percentage PASI 75 responders and were defined as participants achieving ≥ 75% improvement at Week 4
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 300 mg | Ustekinumab
Number analyzed (Participants) | 334 | 335
percentage of participants | 49.7 | 20.6

3. Secondary Outcome: Percentage of Participants With Moderate to Severe Plaque Psoriasis Who Achieved Psoriasis Area and Severity Index (PASI) 90 at Week 52
Description: Psoriasis Area and Severity Index (PASI) is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
  PASI 90 responders were defined as participants achieving ≥ 90% improvement at Week 52
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 300 mg | Ustekinumab
Number analyzed (Participants) | 334 | 335
percentage of participants | 74.9 | 60.6

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Arm/Group | AIN457 300 mg | Ustekinumab
Serious Adverse Events (participants affected / at risk) | 41/335 | 32/336
Other Adverse Events (participants affected / at risk) | 270/335 | 246/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=335) | Ustekinumab (N=336)
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
HAMARTOMA (Congenital, familial and genetic disorders) | 0 | 1
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 | 0
OCULAR HYPERTENSION (Eye disorders) | 1 | 0
VITREOUS ADHESIONS (Eye disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1
DEATH (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
CIRRHOSIS ALCOHOLIC (Hepatobiliary disorders) | 1 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC FATTY LIVER (Hepatobiliary disorders) | 1 | 0
ABSCESS (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
LARYNGITIS (Infections and infestations) | 1 | 0
NASAL ABSCESS (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SCROTAL ABSCESS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1
TONSILLITIS (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INJECTION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRAIN NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
FIBROADENOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
AMNESIA (Nervous system disorders) | 1 | 0
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
FACIAL PARESIS (Nervous system disorders) | 1 | 0
FACIAL SPASM (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0
POSTICTAL PARALYSIS (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LICHENIFICATION (Skin and subcutaneous tissue disorders) | 1 | 0
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 | 1
SEGMENTED HYALINISING VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
VARICOSE VEIN (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=335) | Ustekinumab (N=336)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 12 | 6
DIARRHOEA (Gastrointestinal disorders) | 22 | 24
DYSPEPSIA (Gastrointestinal disorders) | 10 | 9
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 7 | 3
NAUSEA (Gastrointestinal disorders) | 12 | 10
TOOTHACHE (Gastrointestinal disorders) | 12 | 10
VOMITING (Gastrointestinal disorders) | 15 | 7
FATIGUE (General disorders) | 20 | 12
PYREXIA (General disorders) | 14 | 8
BRONCHITIS (Infections and infestations) | 20 | 14
CONJUNCTIVITIS (Infections and infestations) | 18 | 8
CYSTITIS (Infections and infestations) | 9 | 6
EAR INFECTION (Infections and infestations) | 9 | 2
FOLLICULITIS (Infections and infestations) | 11 | 4
GASTROENTERITIS (Infections and infestations) | 11 | 12
HERPES ZOSTER (Infections and infestations) | 1 | 10
INFLUENZA (Infections and infestations) | 33 | 16
NASOPHARYNGITIS (Infections and infestations) | 96 | 87
ORAL CANDIDIASIS (Infections and infestations) | 14 | 2
ORAL HERPES (Infections and infestations) | 13 | 6
PHARYNGITIS (Infections and infestations) | 10 | 12
RHINITIS (Infections and infestations) | 13 | 12
SINUSITIS (Infections and infestations) | 12 | 9
TINEA PEDIS (Infections and infestations) | 10 | 9
TONSILLITIS (Infections and infestations) | 11 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 42 | 36
URINARY TRACT INFECTION (Infections and infestations) | 15 | 7
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 6
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 7 | 0
CONTUSION (Injury, poisoning and procedural complications) | 7 | 8
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 6 | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 36 | 33
BACK PAIN (Musculoskeletal and connective tissue disorders) | 29 | 26
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 9 | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 8 | 6
NECK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 11
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 10 | 11
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
HEADACHE (Nervous system disorders) | 50 | 46
ANXIETY (Psychiatric disorders) | 9 | 3
DEPRESSION (Psychiatric disorders) | 6 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 20
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 32 | 18
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 | 4
ECZEMA (Skin and subcutaneous tissue disorders) | 19 | 12
PRURITUS (Skin and subcutaneous tissue disorders) | 25 | 28
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 8 | 8
PSORIASIS (Skin and subcutaneous tissue disorders) | 22 | 21
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 9 | 5
URTICARIA (Skin and subcutaneous tissue disorders) | 4 | 7
HYPERTENSION (Vascular disorders) | 15 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.